CLINICAL TRIAL: NCT05733572
Title: Safety and Efficacy of Multiple Doses of the PAINLESS Nerve Growth Factor CHF6467 in Paediatric Subjects With Optic Pathway Glioma (OPG). A Randomized Clinical Trial (RCT)
Brief Title: Safety and Efficacy of the PAINLESS Nerve Growth Factor CHF6467 in Optic Pathway Glioma (OPG)
Acronym: NGF-OPG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Benedetto Falsini (Other)
Responsible Party: Sponsor-Investigator, Benedetto Falsini, Professor, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHF6467-OPG
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Optic Pathway Glioma
Keywords: Optic pathway glioma, nerve growth factor; optic atrophy
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Optic Atrophy

STUDY DESIGN:
Intervention Model Description: This is a phase 2a study intended to demonstrate the superiority over placebo of 10 days' treatment with CHF6467 in significantly improving the field of vision of children and young adults with optical pathway glioma, 12 weeks after the start of treatment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: double masking (patients and outcome assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active treatment group (Experimental): active drug treatment group
  Interventions: Drug: CHF6467
- placebo group (Placebo Comparator): pacebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF6467 — drug eyedrops
  Other Names: painless NGF
  Arms: active treatment group
Drug: Placebo — placebo eyedrops
  Arms: placebo group

SUMMARY:
Infantile optic pathway glioma (OPG) is generally benign and slow-growing, but due to infiltration and compression of sensitive neuronal structures in the optical pathways, progressive visual loss is a frequent and highly debilitating complication of the condition. Recently, therapeutic strategies aimed at neuroprotection in the visual pathway rather than reducing the size of the tumor have been studied.

Nerve growth factor (NGF) is a neurotrophin that acts on peripheral and central neurons by binding with high affinity to the trkANGFR receptor, which has tyrosine kinase activity, and with low affinity to the non-selective pan-neurotrophin receptor p75NTR that regulates signaling through trkANGFR. The effect of NGF on target cells depends on the ratio of these two co-distributed receptors on the cell surface.

Recently, two studies have shown that murine NGF can prevent progression of visual damage in OPG patients. These successful exploratory studies (the last of which was a randomized, double-blind, placebo-controlled study) represent a significant reference point in the field of vision loss in OPG patients and provide the basis and rationale for this study using a recombinant form of mutated NGF, painless NGF (CHF6467), which is anticipated to prove devoid of adverse effects related to pain at therapeutic doses.

The purpose of this randomised study is to assess the safety and efficacy of multiple doses of painless NGF CHF6467 eye drops on the visual function of children or young adults with optic pathway gliomas, whether or not associated with type 1 neurofibromatosis. This study will include serial assessments of both optical pathway functionality and morphology, using electrophysiological and magnetic resonance imaging (MRI) techniques of the brain. The comparator will be a placebo preparation based on a physiologically balanced salt solution. This comparator has no effect on retinal function and optic nerve, is painless and perfectly tolerated, as reported by numerous clinical studies including that of our group.

DETAILED DESCRIPTION:
Background and study rationale Nerve growth factor (NGF) is a neurotrophin that acts on peripheral and central neurons by binding with high affinity to the trkANGFR receptor, which has tyrosine kinase activity, and with low affinity to the non-selective pan-neurotrophin receptor p75NTR that regulates signaling through trkANGFR. The effect of NGF on target cells depends on the ratio of these two co-distributed receptors on the cell surface .

Based on its biological effects on neuronal and non-neuronal cells, the therapeutic potential of NGF has been demonstrated for neurodegenerative diseases, such as Alzheimer's disease, and for the healing of corneal and skin tissues damaged by chemical, physical, surgical and autoimmune insults. The development of recombinant forms of NGF that have less pain induction activity, while fully preserving its pleiotrophic properties, can provide a successful strategy to ensure clinical benefit to subjects suffering from a number of relevant conditions.

CHF6467 (hNGF P61S R100E; hNGFp), is a recombinant and "painless" form of human NGF. The mutation at arginine R100 in mature NGF is linked to the rare human genetic disease HSAN V (hereditary sensory sensory neuropathy type V). In HSAN V subjects, a mutation in the NGFB gene (exon 3, nt C661T), turns arginine R100 into tryptophan, producing a syndrome of complete loss of pain perception without affecting most neurological functions.

In addition to the pain-related R100E mutation, CHF6467 has a second "tagging" P61S mutation, which replaces the proline residue at position 61 with a serine residue. This does not produce any known physiological effects, but the "labeled" molecules of hNGFP61S can be detected selectively compared to wild-type hNGF using a specific monoclonal antibody called 4GA, which helps product research and development.

In vitro and in vivo data confirm that CHF6467 (Chiesi) maintains NGF-identical neurotrophic and neuroprotective properties in a variety of cellular tests, while showing significantly reduced pain induction activity in vivo. These data provide the basis for the development of this "painless" form of NGF for the treatment of neurological disorders and other conditions.

Pathology of optic pathway glioma in paediatric age Infantile optical pathway glioma (OPG) is generally benign and slow-growing, but due to infiltration and compression of sensitive neuronal structures in the optical pathways, progressive visual loss is a frequent and highly debilitating complication of the condition. Retinal ganglion cells (RGC) are known to be significantly involved in this process, and the retinal nerve fiber layer (RNFL), the most distal region of the afferent visual pathway composed of RGC axon, is considered a structural marker of visual integrity. RNFL thinning has been associated with clinically noticeable vision loss in children with OPG.

Neurofibromatosis type 1 (NF1) is one of the most common hereditary dominant autosomic syndromes that occur in young children, with an incidence of approximately 1:3000. NF1 OPGs commonly occur in young children, most before the age of 7. Patients are at increased risk of developing tumors of the nervous system, and about 10-20% of children with NF1 will develop low-grade OPG that eventually leads to visual impairment and blindness. NF1-OPG can occur anywhere along the optical pathways, but most frequently occurs in the optic nerves and/or chiasma.

To reduce the progression of visual impairment in OPG patients, standard clinical treatments include surgery, radiotherapy, and chemotherapy, aimed at controlling tumor expansion. All these treatments have high risks and low effectiveness. More recently, therapeutic strategies aimed at neuroprotection in the visual pathway rather than reducing the size of the tumor have been studied.

Rational for the use of CHF6467 in optic pathway glioma Unmodified human NGF has previously been proposed and studied as a treatment for neuropathy associated with diabetes and HIV infection, but the discovery that parenteral administration produced frequent adverse effects of local and generalized pain, which limited dose increase, put an end to this line of investigation.

Experimental animal studies have shown that NGF applied to the conjunctiva reaches the retina and optic pathway and the cerebral cortex, demonstrating biological activity in these regions.

Research into the therapeutic potential of NGF continued, using the well-tolerated murine NGF, and clinical studies demonstrated the safety and efficacy of NGF eye drops in patients with corneal ulcers and severe glaucoma . Finally, an ocular preparation of unmodified recombinant human NGF, cenegermin (Oxervate®) was approved in the EU in 2017 for the treatment of neurotrophic keratitis (EMA, 2017).

Recently, two studies have shown that murine NGF can prevent progression of visual damage in OPG patients (Falsini, 2016). These successful exploratory studies (the last of which was a randomized, double-blind, placebo-controlled study) represent a significant reference point in the field of vision loss in OPG patients and provide the basis and rationale for this study using CHF6467, which is anticipated to prove devoid of adverse effects related to pain at therapeutic doses.

Type and design of the study This is a phase 2a study intended to demonstrate the superiority over placebo of 10 days' treatment with CHF6467 in significantly improving the field of vision of children and young adults with optical pathway glioma, 12 weeks after the start of treatment. The study will be conducted under double blind conditions, using a "staggered" design of parallel groups in order to protect the safety of study participants. The "staggered" design consists of the serial enrolment of several cohorts of subjects in which ascending doses of the drug are administered. In our study there will be 4 cohorts of subjects In each of the first 3 cohorts (A, B and C), 4 children will be randomised to receive either CHF6467 (3) or matching placebo (1) eye drops 10 days. The planned dosing levels will be 1 drop of study medication to each affected eye once daily (Cohort A), twice daily (Cohort B) and three times daily (Cohort C). In cohort D, 24 children will be randomised to receive either CHF6467 (18) or matching placebo (6) eye drops three times a day for 10 days. In the end, a total of 27 subjects will have received CHF6467 and 9 subjects placebo (ratio 3:1).

At the end of the 12-week double-blind and placebo-controlled phase, each subject will be offered the opportunity to join an "open label extension phase" of a further 12 weeks where each subject will receive CHF6467 at the dose corresponding to their blind-phase cohort. (1 drop of CHF6467 1 time a day for 10 days for the 4 subjects of Cohort A, 1 drop of CHF6467 twice a day for 10 days for the 4 subjects of Cohort B, 1 drop of CHF6467 three times a day for 10 days for the 28 subjects of Cohort C and D).

Study goals (primary and secondary endpoints) Objectives of the study The purpose of this randomised study is to assess the safety and efficacy of multiple doses of painless NGF CHF6467 eye drops on the visual function of children or young adults with optic pathway gliomas, whether or not associated with type 1 neurofibromatosis This study will include serial assessments of both optical pathway functionality and morphology, using electrophysiological and magnetic resonance imaging (MRI) techniques of the brain.

The comparator will be a placebo preparation based on a physiologically balanced salt solution. This comparator has no effect on retinal function and optic nerve, is painless and perfectly tolerated, as reported by numerous clinical studies including that of our group

ELIGIBILITY:
Inclusion Criteria:

- 1. Paediatric or adult subjects between the ages of 3 and 40 (including extremes).

2. Diagnosis of OPG-induced visual damage, with or without type 1 neurofibromatosis (NF-1) 3. Stable disease with two brain MRI checks, performed at least 6 months before screening.

Exclusion Criteria:

- 1. concomitant ophthalmological disorder that may affect electrophysiological evaluation.

2. radiotherapy or chemotherapy or any other specific antineoplastic treatment within 9 months before entry.

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
visual field | 6 months
  : the largest radius (the largest) of the field of view measured in degrees of visual angle by kinetic perimetry according to Goldmann with the aim V/4e.

SECONDARY OUTCOMES:
visual evoked potentials | 6 months
  electrophysiological visual retinal and cortical responses

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Falsini, MD, Principal Investigator — universita Cattolica del S. Cuore/Fondazione policlinico A. Gemelli, IRCCS
Locations (1):
- Catholic University, Policlinico A. Gemelli (Hospital), Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
After data collection, anonymized data will be shared with other researchers in the field
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 24 months

REFERENCES:
- [Result] Falsini B, Chiaretti A, Rizzo D, Piccardi M, Ruggiero A, Manni L, Soligo M, Dickmann A, Federici M, Salerni A, Timelli L, Guglielmi G, Lazzareschi I, Caldarelli M, Galli-Resta L, Colosimo C, Riccardi R. Nerve growth factor improves visual loss in childhood optic gliomas: a randomized, double-blind, phase II clinical trial. Brain. 2016 Feb;139(Pt 2):404-14. doi: 10.1093/brain/awv366. Epub 2016 Jan 14. PMID 26767384
- [Result] Falsini B, Chiaretti A, Barone G, Piccardi M, Pierri F, Colosimo C, Lazzareschi I, Ruggiero A, Parisi V, Fadda A, Balestrazzi E, Riccardi R. Topical nerve growth factor as a visual rescue strategy in pediatric optic gliomas: a pilot study including electrophysiology. Neurorehabil Neural Repair. 2011 Jul-Aug;25(6):512-20. doi: 10.1177/1545968310397201. Epub 2011 Mar 26. PMID 21444653
- [Result] Chiaretti A, Falsini B, Servidei S, Marangoni D, Pierri F, Riccardi R. Nerve growth factor eye drop administration improves visual function in a patient with optic glioma. Neurorehabil Neural Repair. 2011 May;25(4):386-90. doi: 10.1177/1545968310395601. Epub 2011 Feb 22. PMID 21343523
- [Result] Abed E, Corbo G, Falsini B. Neurotrophin family members as neuroprotectants in retinal degenerations. BioDrugs. 2015 Feb;29(1):1-13. doi: 10.1007/s40259-014-0110-5. PMID 25408174